CLINICAL TRIAL: NCT06040866
Title: Effects of Pain Neuroscience Education or Biomedical Pain Education With Exercise Training in Primary Dysmenorrhea: A Randomized Clinical Trial
Brief Title: Pain Neuroscience Education and Biomedical Pain Education in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-22038
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study was designed as a parallel group randomized clinical trial. In this study, individuals were planned to be randomly assigned to either Pain Neuroscience Education combined with exercise training or Biomedical Pain Education combined with exercise training groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education (Experimental): In addition to the exercise training (stretching and relaxation exercises), which includes stretching and relaxation exercises routinely used in the field of physiotherapy and rehabilitation in primary dysmenorrhea, the patients in the pain neuroscience education arm will be given pain neuroscience education once a week for 2 weeks. Participants in the pain neuroscience education arm will be given pain neuroscience education once a week for 2 weeks after their first menstruation. The training will be repeated with a reminder session at the end of the 2nd menstruation.
  Interventions: Other: Exercise training; Other: Pain neuroscience education
- Biomedical pain education (Active Comparator): In the biomedical pain education arm, in addition to the exercise training (stretching and relaxation exercises) that includes stretching and relaxation exercises routinely applied in the field of physiotherapy and rehabilitation in primary dysmenorrhea, biomedical pain education will be given once a week for 2 weeks. Participants in the biomedical pain education arm will be given biomedical pain education once a week for 2 weeks after their first menstruation. The training will be repeated with a reminder session at the end of the 2nd menstruation.
  Interventions: Other: Exercise training; Other: Biomedical pain education

INTERVENTIONS:
Other: Exercise training — Exercise training will be applied in the non-menstrual period during 2 menstrual cycles as stretching and relaxation exercises. Stretching exercises will include general stretching and specific stretching exercises and will take approximately 20 minutes in total. After the stretching exercises, relaxation exercise will be performed with diaphragmatic breathing for 10 minutes. The exercises will be performed with music accompanied by a physiotherapist once a week, and it will be recommended to do the exercises as a home program for 2 sessions a week.
Other: Pain neuroscience education — Participants in the first research arm will be given pain neuroscience education once a week for 2 weeks after their first menstruation. The training will be repeated with a reminder session at the end of the 2nd menstruation.
  Arms: Pain neuroscience education
Other: Biomedical pain education — Participants in the second research arm will be given biomedical pain education once a week for 2 weeks after their first menstruation. The training will be repeated with a reminder session at the end of the 2nd menstruation.
  Arms: Biomedical pain education

SUMMARY:
The aim of this study was to compare the effects of biomedical pain education and pain neuroscience education, in addition to routine exercise training, on menstrual pain parameters (pain severity and duration, analgesic use), menstrual stress, somatosensory function, pain catastrophizing, pain beliefs, anxiety/depressive symptom level and quality of life in healthy individuals with primary dysmenorrhea.The design of the study is parallel group, randomized study. Individuals will be randomly assigned to one of the pain neuroscience education or biomedical pain education research arms.

In the literature, there is no study comparing the effects of pain neuroscience education and biomedical pain education in primary dysmenorrhea, which is a problem that affects women's lives significantly. It is important to reveal the effects of different pain trainings for effective pain management in primary dysmenorrhea.

DETAILED DESCRIPTION:
The aim of this study was to compare the effects of biomedical pain education and pain neuroscience education, in addition to routine exercise training, on menstrual pain parameters (pain severity and duration, analgesic use), menstrual stress, somatosensory function, pain catastrophizing, pain beliefs, anxiety/depressive symptom level and quality of life in healthy individuals with primary dysmenorrhea. The design of the study is parallel group, randomized study. The study sample consists of healthy individuals aged 18 years and older with primary dysmenorrhea symptoms.

Individuals will be randomly assigned to one of the two research arms. In addition to the exercise training, which includes stretching and relaxation exercises routinely used in the field of physiotherapy and rehabilitation in primary dysmenorrhea, the patients in the first research arm will be given pain neuroscience education once a week for 2 weeks.

In the second research arm, in addition to the exercise training that includes stretching and relaxation exercises routinely applied in the field of physiotherapy and rehabilitation in primary dysmenorrhea, biomedical pain education will be given once a week for 2 weeks.

Participants will be evaluated in terms of descriptive measurements and outcome measures 3 times in total, before the applications, immediately after the end of the application period, and 3 months after the end of the applications. The primary outcome measurement parameter of the study was determined as the Visual Analog Scale (VAS) score, which is used to determine the severity of menstrual pain. Secondary outcome measures are menstrual stress level to be evaluated with the Menstrual Distress Questionnaire, somatosensory function status to be evaluated with the Central Sensitization Inventory, pain catastrophizing state to be evaluated with the Menstrual Pain Specific Pain Catastrophizing Scale, pain beliefs status to be assessed with the Pain Beliefs Questionnaire, anxiety/depressive symptom level to be evaluated with Depression Anxiety Stress Scales-21 (DASS-21), quality of life to be evaluated with World Health Organization Quality of Life Scale-Short Form and perception of change to be evaluated by 5-point likert scale.

Sample size calculation was performed with G*Power version 3.1 based on previous study results. In the one-way hypothesis design, it was determined that a total of 32 individuals, 16 individuals in each group, should be included in the study in order to reach 80% power with the calculated effect size difference Cohen's d=0.9 and α=0.05 type 1 error. Considering that there might be a 20% loss of individuals during the study, it was decided to include a total of 38 individuals in the study.

In the literature, there is no study comparing the effects of pain neuroscience education and biomedical pain education in primary dysmenorrhea, which is a problem that affects women's lives significantly. It is important to reveal the effects of different pain trainings for effective pain management in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with PD by a gynecologist based on the Primary Dysmenorrhea Consensus Guidelines,
* Nulligravid,
* Not having any known disease,
* Regular menstrual cycle (28±7 days),
* Severity of menstrual pain ≥ 4 cm according to VAS in the last 6 months and during the last menstruation,
* 18 years and over,
* Volunteer healthy female individuals who consented to participate in the study, willing to be randomized, will be included.

Exclusion Criteria:

* Pathological pelvic conditions including endometriosis, chronic pelvic inflammatory disease, adenomyosis, polycystic ovary syndrome, endometrial fibroids/polyps or sexually transmitted diseases,
* History of pelvic or abdominal surgery
* Taking antidepressants, anxiolytics or oral contraceptives,
* Receiving alternative treatment in the last year,
* Individuals using an intrauterine contraceptive device will not be included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Severity of menstrual pain | Change in severity of menstrual pain from baseline up to end of 2 menstrual cycles (each cycle is 28± 7 days)
  Visual Analogue Scale (VAS): This scale is a 10cm horizontal line. 0= no pain/meaning no effect, 10= unbearable pain/ experiencing

SECONDARY OUTCOMES:
Menstrual stress level | Change in level of menstrual stress from baseline up to end of 2 menstrual cycles (each cycle is 28± 7 days)
  Menstrual Distress Questionnaire (MDQ): The scale consists of 47 menstrual symptoms and 8 sub-symptom groups. Complaints are scored from 0 to 4. 0=no symptoms, 1=little, 2=moderate, 3=severe, 4=very severe.
Somatosensory function status | Change in status of somatosensory function from baseline up to end of 2 menstrual cycles (each cycle is 28± 7 days)
  Central Sensitization Inventory (CSI): CSI consists of two parts. Part A contains 25 items that assess somatic and emotional health-related symptoms common in Central sensitization-related disorders.
  Each item is graded on a 5-point scale from (0) "never" to (4) "always", with a maximum total score of 100. Higher scores indicate a higher degree of symptomatology. Section B includes 7 diagnoses of central sensitization syndromes (tension headaches/migraine, fibromyalgia, irritable bowel syndrome, restless legs syndrome, temporomandibular joint disorder, chronic fatigue syndrome, and multiple chemical sensitivities) and three additional diagnoses found to be associated with central sensitization ( depression, anxiety/panic attack, and neck injury); Participants were asked, together with the year of diagnosis, "Has any of the following conditions been diagnosed by a doctor?" contains the question.
Menstrual pain catastrophizing state | Change in state of menstrual pain catastrophizing from baseline up to end of 2 menstrual cycles (each cycle is 28± 7 days)
  Pain Catastrophizing Scale: It has 13 items and consists of 3 sub-dimensions (helplessness, magnification and rumination). Questions are scored between 0-4. Subscales are determined by summing the scores of each item, and the total score (between 0 and 52 points) is calculated with the sum of all items. A higher score means a greater degree of catastrophization.
Menstrual pain beliefs status | Change in status of menstrual pain beliefs from baseline up to end of 2 menstrual cycles (each cycle is 28± 7 days)
  Pain Beliefs Questionnaire (PBQ): It contains 12 items related to pain beliefs. PBQ-O is an 8-item subscale, and PBQ-P is a 4-item subscale. Organic beliefs sub-dimension consists of items 1, 2, 3, 5, 7, 8, 10 and 11, and psychological beliefs sub-dimension consists of items 4, 6, 9 and 12. Participants mark the appropriate answer for themselves on a 6-point response scale ranging from "always" to "never".
Anxiety/depressive symptom level | Change in level of anxiety/depressive symptom from baseline up to end of 2 menstrual cycles (each cycle is 28± 7 days)
  Depression Anxiety Stress Scales-21 (DASS-21): It is a valid measure for depression, anxiety, and stress in adults. Each of the three subscales contains 7 items; each is answered from zero (never) to three (always).
  Higher scores indicate greater levels of depression, anxiety, and stress.
Quality of life level | Change in level of quality of life from baseline up to end of 2 menstrual cycles (each cycle is 28± 7 days)
  World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF): 442 / 5.000 Çeviri sonuçları The WHOQOl-BREF is a 26-item self-administered questionnaire and covers 4 dimensions of quality of life (6 items for psychological health, 7 items for physical health, 3 items for social relationships, and 8 items for environmental health). Except for 3 questions targeting pain and discomfort, need for medical treatment, and negative emotions, each question has response categories ranging from 1 to 5, and a high score indicates high quality of life.
Perception of change | Change in menstrual symptoms immediately after the end of 2 menstrual cycles (each cycle is 28± 7 days) and 3 months after the end of the interventions compared with baseline
  5-point likert scale: Individuals' perception of subjective changes in menstrual pain and other menstrual symptoms with interventions will be evaluated. -2= much worse, -1= slightly worse, 0= no change, 1= slightly better, 2= much better. The changes in the menstrual symptoms of the individuals just after the end of the interventions and 3 months after the end of the interventions will be questioned when compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Özgül, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Büşra Nur Erol, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponce-Fuentes F, Cuyul-Vasquez I, Bustos-Medina L, Fuentes J. Effects of pain neuroscience education and rehabilitation following arthroscopic rotator cuff repair. A randomized clinical trial. Physiother Theory Pract. 2023 Sep 2;39(9):1861-1870. doi: 10.1080/09593985.2022.2061394. Epub 2022 Apr 12. PMID 35412432
- [Background] Li X, Hao X, Liu JH, Huang JP. Efficacy of non-pharmacological interventions for primary dysmenorrhoea: a systematic review and Bayesian network meta-analysis. BMJ Evid Based Med. 2024 May 22;29(3):162-170. doi: 10.1136/bmjebm-2023-112434. PMID 38242565
- [Background] Matthewman G, Lee A, Kaur JG, Daley AJ. Physical activity for primary dysmenorrhea: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2018 Sep;219(3):255.e1-255.e20. doi: 10.1016/j.ajog.2018.04.001. Epub 2018 Apr 7. PMID 29630882
- [Background] Wickstrom K, Edelstam G. Minimal clinically important difference for pain on the VAS scale and the relation to quality of life in women with endometriosis. Sex Reprod Healthc. 2017 Oct;13:35-40. doi: 10.1016/j.srhc.2017.05.004. Epub 2017 May 25. PMID 28844356
- [Background] Moos RH. The development of a menstrual distress questionnaire. Psychosom Med. 1968 Nov-Dec;30(6):853-67. doi: 10.1097/00006842-196811000-00006. No abstract available. PMID 5749738
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Edwards LC, Pearce SA, Turner-Stokes L, Jones A. The Pain Beliefs Questionnaire: an investigation of beliefs in the causes and consequences of pain. Pain. 1992 Dec;51(3):267-272. doi: 10.1016/0304-3959(92)90209-T. PMID 1491853
- [Background] The World Health Organization Quality of Life Assessment (WHOQOL): development and general psychometric properties. Soc Sci Med. 1998 Jun;46(12):1569-85. doi: 10.1016/s0277-9536(98)00009-4. PMID 9672396
- [Background] Jaeschke R, Singer J, Guyatt GH. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989 Dec;10(4):407-15. doi: 10.1016/0197-2456(89)90005-6. PMID 2691207
- [Background] Suren M, Okan I, Gokbakan AM, Kaya Z, Erkorkmaz U, Arici S, Karaman S, Kahveci M. Factors associated with the pain catastrophizing scale and validation in a sample of the Turkish population. Turk J Med Sci. 2014;44(1):104-8. doi: 10.3906/sag-1206-67. PMID 25558568
- [Background] Duzce Keles E, Birtane M, Ekuklu G, Kilincer C, Caliyurt O, Tastekin N, Is EE, Ketenci A, Neblett R. Validity and reliability of the Turkish version of the central sensitization inventory. Arch Rheumatol. 2021 Oct 18;36(4):518-526. doi: 10.46497/ArchRheumatol.2022.8665. eCollection 2021 Dec. PMID 35382371
- [Background] Haldeman S. North American Spine Society: failure of the pathology model to predict back pain. Spine (Phila Pa 1976). 1990 Jul;15(7):718-24. No abstract available. PMID 2145646
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273